CLINICAL TRIAL: NCT00908466
Title: A Phase 1, Open-label, Randomized Clinical Study to Assess the Safety, Tolerability and Bioactivity of Intravitreal and Subconjunctival Injection of Sirolimus in Patients With Non-infectious Uveitis
Brief Title: Sirolimus as Therapeutic Approach to Uveitis
Acronym: SAVE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MacuSight, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00028588
Record Dates: First submitted 2009-04-30; First posted 2009-05-25 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-12

CONDITIONS: Uveitis; Intermediate Uveitis; Posterior Uveitis; Panuveitis
Keywords: Non-infectious; Uveitis; Panuveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior; Panuveitis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravitreal Injection (Experimental): Will receive intravitreal injections of sirolimus 352 µg in study eye on Days 0, 60, and 120.
  Interventions: Drug: Sirolimus (rapamycin)
- Subconjunctival Injection (Experimental): Will receive subconjunctival injections of sirolimus 1320 µg in the study eye on Days 0, 60, and 120.
  Interventions: Drug: Sirolimus (rapamycin)

INTERVENTIONS:
Drug: Sirolimus (rapamycin) — Will receive intravitreal injections of sirolimus (rapamycin) 352 µg in study eye on Days 0, 60, and 120.
  Other Names: Rapamycin, Rapamune, Sirolimus
  Arms: Intravitreal Injection
Drug: Sirolimus (rapamycin) — Will receive subconjunctival injections of sirolimus 1320 µg in the study eye on Days 0, 60, and 120.
  Other Names: Rapamycin, Rapamune, Sirolimus
  Arms: Subconjunctival Injection

SUMMARY:
The purpose of this study is to find out about the safety and effectiveness of the study drug, sirolimus, in patients with uveitis and to utilize the potential effectiveness of sirolimus, and yet to avoid the potential complications of systemic use of the drug. In this study, the investigators will administer sirolimus either around (subconjunctival injection) or inside the eye (intravitreal injection). Local administration of sirolimus to the eye is not expected to have effects on the rest of the body. Therefore, it may offer a safer way than the current methods used to control the inflammation caused by non-infectious uveitis.

DETAILED DESCRIPTION:
Uveitis is a condition in which certain parts of your eye become inflamed. The inflammation is usually recurrent. If the inflammation is not treated adequately, permanent damage to the eye and to the vision may occur. The inflammation can be caused by infectious or non infectious causes. The current research is being done to determine the safety and the usefulness of treatment of non-infectious uveitis using a drug called sirolimus.

Current treatment options for uveitis include oral corticosteroids and drugs that weaken the immune system of the body (i.e., immunosuppressant drugs). Treatment using oral corticosteroids, especially for long periods, may cause many undesirable side effects and complications such as high blood sugar, high blood pressure, bone weakness, obesity, stomach ulcers, abnormal hair growth, and increased risks of infection. In addition to that, in some cases, the disease cannot be controlled even with the highest dose of steroids.

Injection of steroids around and inside the eye can be used to control uveitis. However, the inflammation does not always respond to such kind of treatment. The eyes may develop high pressure and cataract with injections of steroids into the eyes or around the eyes.

On the other hand, despite their potential effectiveness, treatment with drugs that weaken the immune system may cause severe side effects. Increased risk of infection is a common side effect of all the immunosuppressant drugs. The immune system protects the body from infections. When the immune system is suppressed, infections are more likely to happen. Some of these infections are potentially dangerous. Because the immune system protects the body against some forms of cancer, immunosuppressant drugs are also associated with a slightly increased risk of cancer. For example, long-term use of immunosuppressant drugs may carry an increased risk of developing skin cancer as a result of the combination of the drugs and exposure to sunlight. The immunosuppressive drugs are very powerful and can cause serious side effects such as high blood pressure, kidney problems, and liver problems. Some side effects may not show up until years after the medicine is used.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females greater than or equal to 18 years of age;
2. Able to give informed consent and attend all study visits;
3. Have diagnosis of uveitis determined by the Investigator to be non infectious;

   * Have active uveitis, defined as having at least 1+ Vitreous Haze and/or at least 1+ Vitreous Cell Count (SUN scale), and:

     * are receiving no other treatment; or,
     * are receiving prednisone ≥10 mg/day (or equivalent dose of another corticosteroid) and/or at least 1 other systemic immunosuppressant; or, b. Have inactive disease, defined as having 0.5+ Vitreous Haze or less and a grade of 0.5+ Vitreous Cell Count or less (SUN scale), and:
     * are receiving prednisone <10 mg/day (or equivalent dose of another corticosteroid) and/or at least 1 other systemic immunosuppressant.
4. Have posterior, intermediate, or panuveitis; for panuveitis, if an anterior component is present, it must be less than the posterior component;
5. Sufficient inflammation to require systemic treatment and, based on the Investigator's decision, warrants intravitreal or subconjunctival treatment;
6. Best-corrected (ETDRS) visual acuity of 20/40 to 20/400 (approximately 70 to 20 letters) in the study eye;
7. Best- corrected ETDRS visual acuity of 20/400 or better in the fellow eye (approximately 20 letters).

Exclusion Criteria:

1. Patients with bilateral uveitis who are receiving systemic immunosuppressive therapy (e.g., methotrexate, cyclosporine, cyclophosphamide, chlorambucil, mycophenolate mofetil, tacrolimus, or azathioprine) other than prednisone or other corticosteroids for the treatment of the uveitis, and the uveitis in the fellow eyes, in the opinion of the investigator, cannot be controlled with standard local therapies alone;
2. Any significant ocular disease that could compromise vision in the study eye. These include, but are not limited to:

   * Diabetic retinopathy: proliferative diabetic retinopathy (PDR) or non-proliferative diabetic retinopathy (NPDR) that compromise the vision.
   * Age-related macular degeneration;
   * Myopic degeneration with active subfoveal choroidal neovascularization.
3. Any of the following treatments within 90 days prior to Day 0 or anticipated use of any of the following treatments to the study eye:

   * Intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors);
   * Posterior subtenon's steroids.
4. Intraocular surgery within 90 days prior to Day 0 in the study eye;
5. Capsulotomy within 30 days prior to Day 0 in the study eye;
6. If the patient has had glaucoma surgery (trabeculectomy or aqueous shunt device), there must be adequate conjunctiva
7. History of vitreoretinal surgery or scleral buckling
8. Any ocular surgery (including cataract extraction or capsulotomy) of the study eye anticipated within the first 180 days following Day 0;
9. Intraocular pressure ≥25 mmHg in the study eye (glaucoma patients maintained on no more than 2 topical medications with intraocular pressure (IOP) <25 mmHg are allowed to participate);
10. Pupillary dilation inadequate for quality stereoscopic fundus photography in the study eye;
11. Media opacity that would limit clinical visualization;
12. Presence of any form of ocular malignancy in the study eye, including choroidal melanoma;
13. History of herpetic infection in the study eye or adnexa;
14. Presence of known active or inactive toxoplasmosis in either eye;
15. Ocular or periocular infection in either eye;
16. Participation in other investigational drug or device clinical trials within 30 days prior to Day 0, or planning to participate in other investigational drug or device clinical trials within 180 days following Day 0. This includes both ocular and non-ocular clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Vigil EM, Sepah YJ, Watters AL, Sadiq MA, Ansari M, Bittencourt MG, Ibrahim MA, Do DV, Nguyen QD. Assessment of changes in quality of life among patients in the SAVE Study - Sirolimus as therapeutic Approach to uVEitis: a randomized study to assess the safety and bioactivity of intravitreal and subconjunctival injections of sirolimus in patients with non-infectious uveitis. J Ophthalmic Inflamm Infect. 2015 Apr 18;5:13. doi: 10.1186/s12348-015-0044-1. eCollection 2015. PMID 25918559

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravitreal Injection | Subconjunctival Injection
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravitreal Injection | Subconjunctival Injection | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (19.8) | 48 (18.2) | 47 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 6 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 2-step Decrease in Vitreous Haze (VH)
Description: Vitreous Haze is calculated using a 9 step photographic haze in uveitis patients using fundus photograph
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Intravitreal Injection | Subconjunctival Injection
Number analyzed (Participants) | 15 | 15
participants | 4 | 4

2. Secondary Outcome: Change From Baseline VA by ETDRS
Time Frame: 6 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Intravitreal Injection | Subconjunctival Injection
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Injection (N=15) | Subconjunctival Injection (N=15)
Serious Ocular Adverse Event (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal Injection (N=15) | Subconjunctival Injection (N=15)
Inflammation at the injection site (Eye disorders) | 0 (0) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No